CLINICAL TRIAL: NCT03952299
Title: Oxybutynin for Post-surgical Bladder Pain and Urgency
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1336293
Record Dates: First submitted 2019-04-29; First posted 2019-05-16 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Overactive Bladder Syndrome; Neuropathic Bladder
Keywords: Transdermal Oxybutynin
MeSH Terms: conditions — Urinary Bladder, Neurogenic | interventions — Tolterodine Tartrate; oxybutynin

STUDY DESIGN:
Intervention Model Description: Group A: Oral Administration Current standard treatment at U.C. Davis Children's Hospital Oral oxybutynin (5mg) is administered in the preoperative area prior to surgery. Our current regimen is to mix the oxybutynin with the standard preoperative Versed so children do not have to take two dosages.
  Post-operatively oral oxybutynin (5mg) is administered every 8 hours in the hospital.
  Group B: Transdermal Administration Guardian will be given the transdermal patch (3.9mg oxybutynin) at the preoperative appointment with instructions to apply the day prior to surgery. While in the hospital no oral oxybutynin will be prescribed.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oral administration (Active Comparator): Oral oxybutynin (5mg) is administered in the preoperative area prior to surgery. The current regimen is to mix the oxybutynin with the standard preoperative Versed so children do not have to take two dosages.
  Post-operatively oral oxybutynin (5mg) is administered every 8 hours in the hospital.
  Interventions: Drug: Oral Oxybutynin
- Transdermal administration (Experimental): Guardian will be given the transdermal patch (3.9mg oxybutynin) at the preoperative appointment with instructions to apply the day prior to surgery. While in the hospital no oral oxybutynin will be prescribed.
  Interventions: Drug: Oxybutynin Transdermal Patch

INTERVENTIONS:
Drug: Oxybutynin Transdermal Patch — Transdermal patch of oxybutynin will be used instead of oral oxybutynin.
  Other Names: Ditropan XL
  Arms: Transdermal administration
Drug: Oral Oxybutynin — Oral administration of oxybutynin (5mg) every 8 hours in the hospital.
  Other Names: Ditropan XL
  Arms: Oral administration

SUMMARY:
Bladder pain and urgency are common after bladder surgery. The objective is to determine if transdermal administration is superior to oral administration in alleviating pain and urgency.

DETAILED DESCRIPTION:
Pain after bladder surgery is typically controlled with narcotics, non-steroidal anti-inflammatory medications, acetaminophen, regional anesthesia (caudal or epidural) and/or bladder muscle (detrusor) antispasmodic medication. It is often difficult to distinguish bladder pain from a sensation of urinary urgency and most likely patients are experiencing both sensations despite the bladder being empty from the indwelling catheter.

Prior studies on adults have demonstrated the efficacy of preoperative oxybutynin and other antimuscarinics on decreasing catheter-related bladder discomfort in the postoperative period. For pediatric bladder surgery very few studies have been published. Intravenous ketorolac, epidural and caudal analgesia and intravesical ropivacaine have been shown to decrease postoperative bladder spasms. Intravesical oxybutynin has been used in the operating room in adults to decrease post-operative ureteral stent pain.

For open bladder surgery the current pain management standard is intra- and postoperative ketorolac (Q6hrs) and acetaminophen and narcotic as needed. Oral oxybutynin is started pre-operatively and then continued post-operatively every 8 hours. Unfortunately, the bioavailability of oral oxybutynin is poor due to first pass (liver) metabolism of the absorbed medication and a subsequent high level of desethyloxybutynin (DEO) produced by the liver. DEO, responsible for most of the side effects such as dry mouth, dizziness, over-heating, drowsiness and constipation. This metabolite and side effects are less with the transdermal route.

A prior retrospective analysis of children by the investigators did not show a difference in pain between starting oral oxybutynin pre-operatively or initiating medication post-operatively. Whether this was due to no difference, insufficient patient numbers or inability to distinguish bladder spasms from pain is unknown. That study employed the Wong-Baker-Facies scale for pain measurement in children. At the time of that study there was no valid scale for objective measurement of bladder urgency in adults or children. Over the last five years the investigators have developed a validated scale (IRB 647657, 638967) that will allow for a better measure and distinguish bladder and incisional pain from bladder spasms/urgency.

The objective is to determine if transdermal administration is superior to oral administration in alleviating pain and urgency after bladder surgery in children. Oral oxybutynin is a commonly used treatment in children with neuropathic bladder dysfunction and for adults with overactive bladder (OAB) and incontinence. As mentioned, transdermal administration has higher bioavailability and a lower adverse event profile. Transdermal administration has been shown to be safe and efficacious in children with neuropathic bladder disease. The hypothesis is that the transdermal route will decrease bladder pain and urgency if applied prior to surgery with a lower side effect profile.

Based upon the power analysis by Blythe Durbin-Johnson, Ph. D. The investigators plan to evaluate up to 100 patients with early termination if endpoints are reached before 100 subjects.

Outcomes will be compared between groups using two-sample t-tests if the outcome is sufficiently normally distributed, and Wilcoxon-rank sum tests otherwise. With 60 subjects divided among two groups, the two-sample t-test will have 80% power to detect a 0.74 standard deviation difference in outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo bladder surgery that requires an indwelling bladder catheter after surgery.
* Age Range: Four to 8 years of age are eligible for the study.

Exclusion Criteria:

* Patients who have had prior bladder surgery.
* Patients who have neurologic disease that could impair bladder sensation.
* Patients who are already taking antimuscarinic or antispasmodic medications.
* Patients with glaucoma, any neurologic disease, dementia, impaired mentation or disorder of the central nervous system.
* Patients taking any medication that affects the central nervous system such as antidepressant, anxiolytic or antipsychotic medications.
* Less than four years of age cannot have the transdermal patch due to fixed dose. Over 8 years of age: less than 5% of our patients, who undergo this surgery, are over 8 years of age and is usually a rare adolescent. Data in an older cohort may confuse the results since they respond differently to bladder surgery due to larger incision and longer hospital stay with a catheter.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Urgency Scores | Preoperative (one week to two months) to postoperative period (six weeks).
  Mean and peak urgency scores measured using the Pictorial Scale of Bladder Urgency. Children will choose one of four illustrations depicting bladder urgency. These illustrations have been assigned a number 1 through 4. The score of 1 indicates less urgency and a score of 4 indicating greatest urgency.
Pain Scores | Preoperative (one week to two months) to postoperative period (six weeks).
  Mean and peak pain scores assessed using current standard University of California, Davis Medical Center protocols in the preoperative and postoperative period. Depending upon the age of the child and development, the Wong-Baker-Facies scale or numerical scale will be utilized in the hospital, both scored on a scale from 0 to 10, with higher scores indicating greater pain.
Narcotic Usage | Postoperative (six weeks)
  Narcotic usage will be assessed. Morphine and hydrocodone in mg/kg will be recorded and evaluated over the hospitalization period.

CONTACTS AND LOCATIONS:
Overall Officials: Eric A Kurzrock, MD, Principal Investigator — UC Davis Health Center
Locations (1):
- University of California Davis Medical Center (UCDMC), Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chamie K, Chi A, Hu B, Keegan KA, Kurzrock EA. Contemporary open ureteral reimplantation without morphine: assessment of pain and outcomes. J Urol. 2009 Sep;182(3):1147-51. doi: 10.1016/j.juro.2009.05.054. Epub 2009 Jul 22. PMID 19625056
- [Result] Kurzrock EA, Chan YY, Durbin-Johnson BP, DeCristoforo L. Pictorial Urgency Scale: A New Tool for Evaluating Bladder Urgency in Children. J Urol. 2019 Mar;201(3):620-625. doi: 10.1016/j.juro.2018.09.047. PMID 30266334
- [Result] Cartwright PC, Coplen DE, Kogan BA, Volinn W, Finan E, Hoel G. Efficacy and safety of transdermal and oral oxybutynin in children with neurogenic detrusor overactivity. J Urol. 2009 Oct;182(4):1548-54. doi: 10.1016/j.juro.2009.06.058. Epub 2009 Aug 15. PMID 19683731
- [Result] Gleason JM, Daniels C, Williams K, Varghese A, Koyle MA, Bagli DJ, Pippi Salle JL, Lorenzo AJ. Single center experience with oxybutynin transdermal system (patch) for management of symptoms related to non-neuropathic overactive bladder in children: an attractive, well tolerated alternative form of administration. J Pediatr Urol. 2014 Aug;10(4):753-7. doi: 10.1016/j.jpurol.2013.12.017. Epub 2014 Jan 17. PMID 24477421
- See also: Learn more or sign up for the study here! — https://studypages.com/s/a-study-of-oral-vs-transdermal-through-skin-patch-oxybutynin-for-post-surgical-bladder-pain-and-urgency-in-children-201477/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-09): https://cdn.clinicaltrials.gov/large-docs/99/NCT03952299/Prot_SAP_002.pdf
  • Informed Consent Form (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/99/NCT03952299/ICF_000.pdf